CLINICAL TRIAL: NCT04323709
Title: Levosimendan for Reducing Veno-arterial ECMO Weaning Failure During Refractory Cardiogenic Shock: a Retrospective Propensity Score Analysis
Brief Title: Levosimendan for Veno-arterial ECMO Weaning
Acronym: WEANECMO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: WEANECMO_2020
Record Dates: First submitted 2020-03-06; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Cardiogenic Shock; Refractory Shock
Keywords: Refractory cardiogenic shock; Levosimendan; VA-ECMO (Veno-Arterial ExtraCorporeal Membrane Oxygenation)
MeSH Terms: conditions — Shock, Cardiogenic; Shock | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- levosimendan group: All patients undergoing VA-ECMO from January 2012 to December 2018 and treated with levosimendan were eligible.
  Interventions: Other: Data collection; Other: Data analysis
- group control: All patients undergoing VA-ECMO from January 2012 to December 2018 but not treated with levosimendan were eligible.
  Interventions: Other: Data collection; Other: Data analysis

INTERVENTIONS:
Other: Data collection — Clinical data are collected from the medical record of the institution. At admission, date were collected on age, gender, body mass index, Simplified Acute Physiology Score II, Sequential Organ Failure Assessment, hypertension, diabetes, hypercholesterolemia, smoking, history of stroke or congestive heart failure, coronary or peripheral artery disease, renal failure with dialysis, Left Ventricular Ejection Fraction(LVEF), Tricuspid Annular Plane Systolic Excursion, mean arterial pressure, heart rate, central venous pressure, ScvO2, presence of an intra-aortic balloon pump and biochemical parameters. During hospitalization data were collected on reason for initiation of VA-ECMO and its characteristics (duration, type, flow L/min, RPM, FiO2), length of stay in ICU, catecholamines and inotropes maximal dose and length of administration, patients with heart transplantation or LVAD. In patients with levosimendan treatment, timing of administration regarding ECMO canulation was collected
Other: Data analysis — Continuous variables were presented as mean ± standard deviation and compared using Student's t-test or Mann-Whitney U-test depending on their normality. Categorical variables were presented as counts and percentages and compared using Pearson's chi-squared test or Fisher's exact test, as appropriate. Survival at day 28 was estimated using the Kaplan-Meier method and compared using the log rank test. Investigators conducted a multivariable logistic regression with propensity score matching, which was defined as the probability of exposure to levosimendan. Results were reported as odd ratios (ORs) together its 95%CI assuming a 5% level of statistical significance. All analyses were carried out using STATA 15.0 (Stata Corp, College Station, Texas 77845 USA).

SUMMARY:
Veno-arterial extracorporeal membrane oxygenation (VA-ECMO) is a temporary mechanical circulatory support that has been increasingly used over the last decade to restore and maintain adequate end-organ perfusion, with data suggesting improvement in outcome for patients with refractory cardiogenic shock. Nevertheless, VA-ECMO weaning should be questioned every day during patient's support. Indeed, studies have shown that the incidence of severe complications related to ECMO is associated with longer circulatory support duration. Inotropes such as dobutamine are currently used to improve myocardial contractility during VA-ECMO support with the aim to enhance left ventricular ejection, aortic valve opening and to shorten ECMO duration. However, many data suggest an increase in mortality related to predisposition to myocardial ischemia and arrythmias. Levosimendan is a calcium sensitizing inotropic agent with systemic, coronary and pulmonary vasodilatory properties and specific cardioprotective effect without increasing myocardial oxygen consumption. The use of levosimendan in patients undergoing VA-ECMO may therefore be of interest both to reduce the duration of mechanical support and to minimize severe complication with few data suggesting a potential benefit of levosimendan for VA-ECMO weaning and survival in post-cardiotomy low cardiac output syndrome with improvement of endothelial function and hemodynamics. Investigators therefore sought to investigate whether the use of levosimendan improves weaning for patients undergoing VA-ECMO support for refractory cardiogenic shock hospitalized in the surgical intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* All consecutive patients admitted with VA-ECMO support for refractory cardiogenic shock
* All consecutive patients admitted for lobectomy or wedge video-assisted thoracoscopy
* Levosimendan administration was left to the discretion of the attending clinician

Exclusion Criteria:

* Age < 18 years
* VA-ECMO duration < 48h
* VA-ECMO for refractory cardiac arrest
* Right heart or veno-venous ECMO
* VA-ECMO for circulatory failure following lung transplant surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators performed a retrospective single-center cohort study. All patients undergoing VA-ECMO from January 2012 to December 2018 were eligible and divided into two groups: group levosimendan and group control (without levosimendan
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
VA-ECMO weaning failure defined as death | 24 hours
  The primary endpoint was VA-ECMO weaning failure defined as death during ECMO support or death within 24h after ECMO removal.

SECONDARY OUTCOMES:
Impact of exposure to levosimendan (at day 28) | Day 28
  Secondary endpoints were the impact of exposure to levosimendan on mortality at day 28 after VA-ECMO canulation.
Impact of exposure to levosimendan (at 6 months) | 6 months
  Secondary endpoints were the impact of exposure to levosimendan on mortality at 6 months after VA-ECMO canulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France

REFERENCES:
- [Derived] Guilherme E, Jacquet-Lagreze M, Pozzi M, Achana F, Armoiry X, Fellahi JL. Can levosimendan reduce ECMO weaning failure in cardiogenic shock?: a cohort study with propensity score analysis. Crit Care. 2020 Jul 16;24(1):442. doi: 10.1186/s13054-020-03122-y. PMID 32677985